CLINICAL TRIAL: NCT04925687
Title: Phase 1 Study of the Feasibility and Safety of Intravitreal Autologous Bone Marrow CD34+ Stem Cell Therapy for Eyes With Vision Loss From Retinitis Pigmentosa
Brief Title: Phase 1 Study of Intravitreal Autologous CD34+ Stem Cell Therapy for Retinitis Pigmentosa
Acronym: BMSCRP1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Cures Within Reach (Other); The Retina Society (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1743714
Record Dates: First submitted 2021-06-02; First posted 2021-06-14 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; stem cell; retinal degeneration; intravitreal
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravitreal autologous CD34+ cells (Experimental): Intravitreal injection of autologous CD34+ cells harvested from bone marrow under GMP conditions
  Interventions: Biological: Intravitreal autologous CD34+ cells

INTERVENTIONS:
Biological: Intravitreal autologous CD34+ cells — Autologous CD34+ cells harvested from bone marrow injected intravitreal

SUMMARY:
In this Phase 1 open-labeled prospective study, one eye of each participant with vision loss from retinitis pigmentosa will be administered intravitreal injection of autologous CD34+ stem cells harvested from bone marrow. Each participant will be examined serially for 6 months after study injection to determine safety and feasibility of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age 2. Visual Acuity at Presentation of 20/100 to Counting Fingers or constriction of peripheral visual field 360 degrees to <10 degrees by perimetry if BCVA is better than 20/100, duration of vision loss > 3 months 3. Vision loss due to retinitis pigmentosa 4. The study eye has the worse visual acuity or peripheral constriction. 14. Able and willing to sign consent 15. Able to keep follow-up appointments for at least 6 months

Exclusion Criteria:

1. Other concurrent optic nerve or retinal disease in study eye affecting vision
2. History of active retinal or choroidal neovascularization or macular edema in study eye requiring on-going intravitreal or periocular therapy in study eye
3. Active eye or systemic infection
4. Significant media opacity in the study eye precluding view of the fundus for examination, photography or optical coherence tomography (OCT)

9. Other cause for vision loss in the study eye 10. History of coagulopathy or other hematologic abnormality 11. Use of coumadin within 3 days of enrollment 12. Concurrent immunosuppressive therapy 13. History of allergy to fluorescein dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Safety of intravitreal injection of autologous CD34+ cells | 6 months
  Number and severity of Ocular and systemic adverse events
Feasibility of intravitreal injection of autologous CD34+ cells | Baseline
  Number of CD34+ cells harvested for intravitreal injection

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months
  Change in number of letters read in study eye from baseline
Best corrected visual acuity | 1 month
  Change in number of letters read in study eye from baseline
Visual Field | 6 months
  Change in visual field area in study eye from baseline
Visual Field | 1 month
  Change in visual field area in study eye from baseline
Electroretinography | 6 months
  Change in a and b wave amplitude in study eye from baseline
Electroretinography | 1 month
  Change in a and b wave amplitude in study eye from baseline
National Eye Institute Vision Questionnaire | 6 months
  Change in Vision Questionnaire compared to baseline
National Eye Institute Vision Questionnaire | 1 month
  Change in Vision Questionnaire compared to baseline
Microperimetry | 6 months
  Change in average threshold from baseline
Microperimetry | 6 months
  Change percent reduced sensitivity from baseline
Microperimetry | 1 month
  Change in average threshold from baseline
Microperimetry | 1 month
  Change in percent reduced sensitivity from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Park, MD PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No